CLINICAL TRIAL: NCT02697136
Title: Phase 3, Multicenter, Randomized, 48 Week, Double Blind, Parallel Group, Placebo Controlled Study to Evaluate Efficacy and Safety of CER-001 on Vessel Wall Area in Patients With Genetically Defined Familial Primary Hypoalphalipoproteinemia
Brief Title: CER-001 Therapy as a Novel Approach to Treat Genetic Orphan Diseases
Acronym: TANGO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Cerenis Therapeutics, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CER-001-CLIN-009
Record Dates: First submitted 2016-02-17; First posted 2016-03-03 (Estimated); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Familial Hypoalphalipoproteinemia
Keywords: Low HDL; Low apoA-I; ABCA-1 mutations; ApoA-I mutations
MeSH Terms: conditions — Hypoalphalipoproteinemias | interventions — CER-001; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CER-001 (Experimental): CER-001 infusion; 9 weekly infusions followed by 20 biweekly infusions
  Interventions: Drug: CER-001
- Placebo (Placebo Comparator): Saline infusion; 9 weekly infusions followed by 20 biweekly infusions
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CER-001 — Recombinant human apoA-I/phospholipid complexes
  Other Names: CAS 138-3435-67-3
  Arms: CER-001
Drug: Placebo — 0.9% Sodium Chloride Injection, USP
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the impact of 29 intravenous infusions of CER-001 vs. placebo, given at weekly (9 infusions) and biweekly (20 infusions) intervals on carotid vessel wall area as measured by 3TMRI, when administered to patients with familial primary hypoalphalipoproteinemia with proven CVD and appropriate background lipid-lowering therapy.

DETAILED DESCRIPTION:
Subjects will be required to have acceptable baseline 3TMRI imaging of carotid arteries. Subjects meeting all eligibility criteria will be randomized to receive CER-001 or placebo (2:1 randomization scheme). Randomized subjects will return weekly for a total of 9 infusions and then biweekly for an additional 20 infusions. 3TMRI imaging of the carotid and femoral arteries will be performed at Week 8, Week 24 (primary endpoint) and Week 48. The total study duration from randomization can range from 50 to 54 weeks for patients completing the study as designed.

ELIGIBILITY:
Main Inclusion Criteria:

* Male and female patients, aged 18 and above.
* ApoA-I < 70 mg/dL
* Symptomatic or asymptomatic cardiovascular disease
* Diagnosis of genetically confirmed HDL-c deficiency due to defects in genes coding for ABCA1 and/or ApoA-1
* Stable doses of lipid lowering therapies for at least 6 weeks prior to baseline procedures

Main Exclusion Criteria:

* Females of childbearing potential
* Patients with LCAT mutations
* Patients who experienced recent cardiovascular or cerebrovascular events
* Hypertriglyceridemia (>500 mg/dL)
* Severe anemia (Hgb < 10 g/dL)
* Uncontrolled diabetes (HbA1c >10%)
* Congestive heart failure (NYHA class II or higher)
* Contraindication for MRI scanning (e.g., implanted metal objects, claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik SG Stroes, MD PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (19):
- Investigative Site, Salt Lake City, Utah, United States
- Investigative Site, La Louvière, Belgium
- Canada (5):
  - Investigative Site, Vancouver, British Columbia
  - Investigative Site, Halifax, Nova Scotia
  - Investigative Site, London, Ontario
  - Investigative Site, Chicoutimi, Quebec
  - Investigative Site, Montreal, Quebec
- France (4):
  - Investigative Site, Lille
  - Investigative Site, Montpellier
  - Investigative Site, Rouen
  - Investigative Site, Toulouse
- Israel (2):
  - Investigative Site, Jerusalem
  - Investigative Site, Tel Aviv
- Italy (4):
  - Investigative Site, Genoa
  - Investigative Site, Milan
  - Investigative Site, Pisa
  - Investigative Site, Rome
- Netherlands (2):
  - Investigative Site, Amsterdam
  - Investigative Site, Utrecht

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CER-001 | Placebo
Started | 20 | 10
Completed Week 8 (Induction Period) | 18 | 10
Completed Week 24 (Maintenance Period) | 17 | 10
Completed (Completed Week 48 (Extension Period)) | 17 | 10
Not Completed | 3 | 0
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CER-001 | Placebo | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Median (Full Range); unit: years] | 54.65 [34.5 to 65.7] | 53.27 [43.5 to 62.1] | 53.79 [34.5 to 65.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 15 | 7 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 3 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 7 | 19
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 3 | 6
  Netherlands | 9 | 6 | 15
  Belgium | 1 | 1 | 2
  United States | 2 | 0 | 2
  Italy | 2 | 0 | 2
  Israel | 1 | 0 | 1
  France | 2 | 0 | 2
Mutation [Count of Participants; unit: Participants]
  ApoA-I Mutation Only | 8 | 4 | 12
  ABCA1 Mutation Only | 11 | 5 | 16
  ApoA-I and ABCA1 Mutations | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Vessel Wall Area (MVWA) of the Carotid Artery
Description: Change from baseline to Week 24 carotid MVWA; CER-001 versus placebo; measured by 3TMRI
Time Frame: Baseline to Week 24
Population: Modified Intent-to-Treat -- All patients randomized to treatment who have baseline and Week 24 carotid 3TMRI performed
Measure: Least Squares Mean (95% Confidence Interval); unit: mm2
Arm/Group | CER-001 | Placebo
Number analyzed (Participants) | 17 | 10
mm2 | -0.3 [-1.0 to 0.4] | 0.5 [-0.4 to 1.4]
Statistical Analysis 1: Comparison: CER-001 vs Placebo; Test type: Other — Linear mixed model to test for superiority and non-inferiority. Equivalence was defined as a difference of less than 6.7% in MVWA, based on a pilot study. Using an assumed standard deviation of 4.5% and a 2:1 randomization scheme to maximize exposure to active drug, 16 completing patients in the CER-001 group and 8 in the placebo group (24 total completers for mITT) would yield 90% power to detect a difference from baseline versus placebo of 6.7%, using two-tailed testing with α=0.05; p = 0.185, Mixed Models Analysis; Difference in LS Means = -0.08, 95% CI 2-sided [-1.9 to 0.4]

2. Secondary Outcome: Change in Mean Vessel Wall Area (MVWA) of the Carotid Artery
Description: Change from baseline to Week 8 carotid MVWA; CER-001 versus placebo; measured by 3TMRI
Time Frame: Baseline to Week 8
Population: Modified Intent-to-Treat -- All patients randomized to treatment who have baseline and Week 8 carotid 3TMRI performed
Measure: Least Squares Mean (95% Confidence Interval); unit: mm2
Arm/Group | CER-001 | Placebo
Number analyzed (Participants) | 16 | 10
mm2 | 0.2 [-0.5 to 0.9] | -0.5 [-1.4 to 0.4]
Statistical Analysis 1: Comparison: CER-001 vs Placebo; Test type: Other — Linear mixed model to test for superiority and non-inferiority. Equivalence was defined as a difference of less than 6.7% in MVWA, based on a pilot study; p = 0.217, Mixed Models Analysis; Difference in LS Means = 0.7, 95% CI 2-sided [-0.4 to 1.8]

3. Secondary Outcome: Change in Mean Vessel Wall Area (MVWA) of the Carotid Artery
Description: Change from baseline to Week 48 carotid MVWA; CER-001 versus placebo; measured by 3TMRI
Time Frame: Baseline to Week 48
Population: Modified Intent-to-Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: mm2
Arm/Group | CER-001 | Placebo
Number analyzed (Participants) | 15 | 9
mm2 | -0.1 [-1.0 to 0.8] | 0.1 [-1.1 to 1.3]
Statistical Analysis 1: Comparison: CER-001 vs Placebo; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.832, Mixed Models Analysis; Difference in LS Means = -0.2, 95% CI 2-sided [-1.6 to 1.3]

4. Secondary Outcome: Change in Target to Background Ratio (TBR) of the Carotid Artery
Description: Change from baseline to Week 24 in carotid TBR; CER-001 versus placebo; measured by FDG-PET
Time Frame: Baseline to Week 24
Population: Carotid MRIs were analyzed for TBR in very few patients. Carotid imaging was performed for during the study, but the images were not read, measured or analyzed for TBR by the central imaging lab following termination of the study and closure of the Sponsor company (Cerenis Therapeutics). No funds were made available by the company's Board of Directors to complete these activities. At that time, paired data (baseline and 24 week) was available for only five patients.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | CER-001 | Placebo
Number analyzed (Participants) | 4 | 1
Ratio | 0.30 (0.160) | 0.35 (0.215)

5. Other Pre Specified Outcome: Change in Femoral MVWA
Description: Assessed by 3TMRI; change from baseline; CER-001 versus placebo
Time Frame: Baseline, Weeks 8, 24 and 48
Population: Femoral imaging was performed for some patients during the study, but the images were not read, measured or analyzed for Mean Vessel Wall Area by the central imaging lab following termination of the study and closure of the Sponsor company (Cerenis Therapeutics). No funds were made available by the company's Board of Directors to complete these activities.
Arm/Group | CER-001 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year (48 weeks of double-blind treatment plus 4 weeks of post-treatment follow-up) for subjects opting out of open-label safety extension. 18 months (48 weeks of double-blind treatment followed by 26-week open-label CER-001 treatment plus 4 weeks of post-treatment follow-up) for subjects opting into open-label safety extension.
Description: Adverse events were collected by querying subjects at each study visit (weekly through Week 8, biweekly from Week 10 to 48 [end of therapy], at Week 52 [4 weeks post-therapy]). During the open-label extension, adverse events were collected biweekly from Weeks 50 through 78. Physical exams and clinical laboratory sampling to determine any adverse changes from baseline were performed at Weeks 4, 8, 16, 24, 32, 40, 48 (end of therapy) and 52 (4 weeks post-therapy).
Groups:
- CER-001 DB Treatment: CER-001 infusion; 9 weekly infusions followed by 20 biweekly infusions plus 12 biweekly infusions during the optional OL extension
  CER-001: Recombinant human apoA-I/phospholipid complexes
- Placebo DB Treatment: Saline infusion; 9 weekly infusions followed by 20 biweekly infusions
  Placebo: 0.9% Sodium Chloride Injection, USP
- CER-001 OL Treatment: 12 biweekly infusions during the optional OL extension
  CER-001: Recombinant human apoA-I/phospholipid complexes
Arm/Group | CER-001 DB Treatment | Placebo DB Treatment | CER-001 OL Treatment
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10 | 0/26
Serious Adverse Events (participants affected / at risk) | 4/20 | 0/10 | 0/26
Other Adverse Events (participants affected / at risk) | 19/20 | 9/10 | 9/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CER-001 DB Treatment (N=20) | Placebo DB Treatment (N=10) | CER-001 OL Treatment (N=26)
Angina Unstable (Cardiac disorders) | 1 (1) | 0 (0) | NA
Vascular Stent Stenosis (General disorders) | 1 (1) | 0 (0) | NA
Complication Associated with Device (General disorders) | 1 (1) | 0 (0) | NA — Coiling of arterial stent
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 (0) | NA
Pyelonephritis Acute (Infections and infestations) | 1 (1) | 0 (0) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CER-001 DB Treatment (N=20) | Placebo DB Treatment (N=10) | CER-001 OL Treatment (N=26)
Nasopharyngitis (Infections and infestations) | 5 | 3 | 2
Hordeolum (Infections and infestations) | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Eye Infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Tooth Infection (Infections and infestations) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Abnormal Faeces (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 0
Faeces Hard (Gastrointestinal disorders) | 0 | 0 | 1
Lip Dry (Gastrointestinal disorders) | 1 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 0
Impaired Healing (General disorders) | 0 | 1 | 0
Influenza Like Illness (General disorders) | 1 | 0 | 0
Infusion Site Bruising (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Peripheral Swelling (General disorders) | 1 | 0 | 0
Pseudoangina (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2
Headache (Nervous system disorders) | 1 | 2 | 0
Aphonia (Nervous system disorders) | 0 | 1 | 0
Balance Disorder (Nervous system disorders) | 0 | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 0
Palpitations (Cardiac disorders) | 2 | 0 | 0
Cartilage Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Albumin Urine Present (Investigations) | 1 | 0 | 0
Heart Rate Irregular (Investigations) | 0 | 0 | 1
Red Blood Cells Urine Positive (Investigations) | 0 | 1 | 0
White Blood Cells Urine Positive (Investigations) | 0 | 1 | 0
Rask (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dental Care (Surgical and medical procedures) | 1 | 0 | 0
Endodontic Procedure (Surgical and medical procedures) | 0 | 1 | 0
Hair Transplant (Surgical and medical procedures) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1
Peripheral Coldness (Vascular disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Lagophthalmos (Eye disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can publish results only 12 months from study completion and database lock or after the multicenter publication, whichever is sooner. All proposed publications/disclosures must be made available for sponsor review 90 days prior to public release and sponsor must respond within 45 days. The sponsor cannot require changes to the communication.

DOCUMENTS (2):
  • Study Protocol (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT02697136/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT02697136/SAP_001.pdf